CLINICAL TRIAL: NCT00096096
Title: A Phase II Study of the Combination of Tacrolimus and Mycophenolate Mofetil for the Prevention of Acute Graft-Versus-Host Disease
Brief Title: Tacrolimus and Mycophenolate Mofetil in Preventing Acute Graft-Versus-Host Disease in Patients With Advanced Hematologic Cancer Who Are Undergoing Donor Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Supportive Care
Other Study IDs: 1893.00; FHCRC-1893.00; CDR0000391026 (Registry Identifier: PDQ)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2010-05-13 (Estimated); Status verified 2010-05

CONDITIONS: Chronic Myeloproliferative Disorders; Graft Versus Host Disease; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: graft versus host disease; accelerated phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; recurrent adult Hodgkin lymphoma; refractory multiple myeloma; recurrent adult Burkitt lymphoma; chronic idiopathic myelofibrosis; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent mantle cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult lymphoblastic lymphoma; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; adult acute lymphoblastic leukemia in remission; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; chronic myelomonocytic leukemia; refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; refractory anemia with ringed sideroblasts; refractory hairy cell leukemia; juvenile myelomonocytic leukemia; chronic eosinophilic leukemia; chronic neutrophilic leukemia; chronic phase chronic myelogenous leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; recurrent/refractory childhood Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; refractory chronic lymphocytic leukemia; refractory cytopenia with multilineage dysplasia; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; adult acute myeloid leukemia in remission; childhood acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); childhood acute lymphoblastic leukemia in remission; childhood chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; myelodysplastic/myeloproliferative disease, unclassifiable; nodal marginal zone B-cell lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; splenic marginal zone lymphoma; atypical chronic myeloid leukemia; stage III childhood large cell lymphoma; stage IV childhood large cell lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; stage III childhood small noncleaved cell lymphoma; stage IV childhood small noncleaved cell lymphoma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Graft vs Host Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Accelerated Phase; Hodgkin Disease; Burkitt Lymphoma; Primary Myelofibrosis; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelomonocytic, Chronic; Anemia, Refractory, with Excess of Blasts; Leukemia, Hairy Cell; Leukemia, Myelomonocytic, Juvenile; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Acute; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Mycosis Fungoides; Sezary Syndrome; Congenital Abnormalities; Blast Crisis; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative | interventions — Mycophenolic Acid; Tacrolimus

INTERVENTIONS:
Drug: mycophenolate mofetil
Drug: tacrolimus

SUMMARY:
RATIONALE: Tacrolimus and mycophenolate mofetil may be an effective treatment for graft-versus-host disease caused by donor stem cell transplantation.

PURPOSE: This phase II trial is studying how well giving tacrolimus together with mycophenolate mofetil works in preventing acute graft-versus-host disease in patients who are undergoing donor stem cell transplantation for advanced hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of tacrolimus and mycophenolate mofetil in preventing acute graft-vs-host disease in patients with advanced hematologic malignancies undergoing allogeneic peripheral blood stem cell transplantation.

Secondary

* Determine the safety of this regimen in these patients.

OUTLINE: This is a non-randomized study.

Patients receive tacrolimus IV continuously or orally twice daily on days -1 to 60 followed by a taper to day 180. Patients also receive mycophenolate mofetil IV over 2 hours or orally twice daily on days 0-60 followed by a taper to day 180. Treatment is discontinued at day 180 in the absence of graft-vs-host disease.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 5-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following hematologic malignancies:

  * Acute myeloid leukemia beyond first complete remission (CR1)
  * Acute lymphoblastic leukemia beyond CR1
  * Chronic myelogenous leukemia in second chronic phase, accelerated phase, or blastic phase
  * Non-Hodgkin's lymphoma beyond CR2
  * Hodgkin's lymphoma beyond CR2
  * Multiple myeloma (any stage)
  * Myelodysplastic syndromes beyond refractory anemia (including chronic myelomonocytic leukemia)
  * Any refractory hematologic malignancy
* Advanced disease
* Scheduled for transplantation of mobilized allogeneic peripheral blood stem cells

  * Genotypically HLA-identical stem cell donor available

PATIENT CHARACTERISTICS:

Age

* 65 and under

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* SGOT and SGPT ≤ 2.0 times ULN

Renal

* Creatinine clearance ≥ 60 mL/min

Pulmonary

* No acute pulmonary infection by chest x-ray
* No severe hypoxemia (partial O_2 < 70% of predicted) AND DLCO < 70% of predicted
* No mild hypoxemia (partial O_2 < 80% of predicted) AND DLCO < 60% of predicted

Other

* Not pregnant or nursing
* Negative pregnancy test
* No active systemic infection not controlled with antimicrobial therapy
* HIV negative (HIV-1 or other virus)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent T-cell depleted hematopoietic stem cell graft

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-08; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Efficacy

SECONDARY OUTCOMES:
Safety
Area under the curve of plasma mycophenolic acid

CONTACTS AND LOCATIONS:
Overall Officials: Richard Nash, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States